CLINICAL TRIAL: NCT04381936
Title: Randomised Evaluation of COVID-19 Therapy
Acronym: RECOVERY
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: UK Research and Innovation (Other); National Institute for Health Research, United Kingdom (Other Government); Wellcome Trust (Other); Bill and Melinda Gates Foundation (Other); Department for International Development, United Kingdom (Other Government); Health Data Research UK (Unknown); Medical Research Council Population Health Research Unit (Unknown); NIHR Health Protection Research Unit in Emerging and Zoonotic Infections (Unknown); Flu Lab (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NDPHRECOVERY; 2020-001113-21 (EudraCT Number); ISRCTN50189673 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2020-05-07; First posted 2020-05-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Severe Acute Respiratory Syndrome
Keywords: COVID-19; SARS-CoV-2; SARS coronavirus 2; SARS; Viral pneumonia syndrome; Community-acquired pneumonia; Bacterial pneumonia syndrome; Influenza A; Influenza B
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Community-Acquired Pneumonia | interventions — Lopinavir; Adrenal Cortex Hormones; Hydroxychloroquine; Azithromycin; tocilizumab; Immunoglobulins; casirivimab and imdevimab drug combination; Aspirin; Colchicine; baricitinib; Interleukin 1 Receptor Antagonist Protein; Dimethyl Fumarate; empagliflozin; sotrovimab; molnupiravir; nirmatrelvir and ritonavir drug combination; baloxavir; Oseltamivir

STUDY DESIGN:
Intervention Model Description: RECOVERY participants are randomly allocated between one or more treatment arms. Not all treatments are available in all countries.
  COVID-19:
  Parts A to D, and the arm for children with PIMS-TS, have been discontinued.
  Part E: randomisation between no additional treatment vs high dose corticosteroids
  Part F: discontinued
  Part J: randomisation between no additional treatment vs sotrovimab
  Part K: discontinued
  Part L: discontinued
  Influenza:
  Part G: randomisation between no additional treatment vrs baloxavir marboxil
  Part H: randomisation between no additional treatment vrs oseltamivir
  Part I: randomisation between no additional treatment vrs Low-dose corticosteroids: Dexamethasone
  Community-acquired pneumonia:
  Part M: randomisation between no additional treatment vrs Low-dose corticosteroids: Dexamethasone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (23):
- Standard Care (No Intervention): Patient receives usual hospital care
- Low dose corticosteroids (Active Comparator): First (main) randomisation part A
  [This arm is now closed to recruitment]
  Interventions: Drug: Corticosteroid
- Hydroxychloroquine (Active Comparator): First (main) randomisation part A
  [This arm is now closed to recruitment]
  Interventions: Drug: Hydroxychloroquine
- Lopinavir-Ritonavir (Active Comparator): First (main) randomisation part A
  [This arm is now closed to recruitment]
  Interventions: Drug: Lopinavir-Ritonavir
- Azithromycin (Active Comparator): First (main) randomisation part A
  [This arm is now closed to recruitment]
  Interventions: Drug: Azithromycin
- Convalescent plasma (Active Comparator): First (main) randomisation part B
  [This arm is now closed to recruitment]
  Interventions: Biological: Convalescent plasma
- Tocilizumab (Active Comparator): Participants with progressive COVID-19 (as evidenced by hypoxia and an inflammatory state) may undergo randomisation between Tocilizumab and no additional treatment.
  (Children with COVID-19 pneumonia are not eligible for this comparison).
  [This arm is now closed to recruitment]
  Interventions: Drug: Tocilizumab
- Intravenous Immunoglobulin (Active Comparator): First (main) randomisation part A (children only)
  [This arm is now closed to recruitment]
  Interventions: Biological: Immunoglobulin
- Synthetic neutralising antibodies (Active Comparator): First (main) randomisation part B.
  [This arm is now closed to recruitment]
  Interventions: Drug: Synthetic neutralising antibodies
- Aspirin (Active Comparator): First (main) randomisation part C
  [This arm is now closed to recruitment]
  Interventions: Drug: Aspirin
- Colchicine (Active Comparator): First (main) randomisation part A
  [This arm is now closed to recruitment]
  Interventions: Drug: Colchicine
- Baricitinib (Active Comparator): First (main) randomisation part D
  [This arm is now closed to recruitment]
  Interventions: Drug: Baricitinib
- Anakinra (Active Comparator): Randomisation for children only with PIMS-TS
  (Children with COVID-19 pneumonia are not eligible for this comparison).
  [This arm is now closed to recruitment]
  Interventions: Drug: Anakinra
- Dimethyl fumarate (Active Comparator): First (main) randomisation part A (UK adults only; early phase assessment)
  [This arm is now closed to recruitment]
  Interventions: Drug: Dimethyl fumarate
- High Dose Corticosteroids (Active Comparator): First (main) randomisation part E
  Interventions: Drug: High Dose Corticosteroid
- Empagliflozin (Active Comparator): First (main) randomisation part F
  [This arm is now closed to recruitment]
  Interventions: Drug: Empagliflozin
- Sotrovimab (Active Comparator): First (main) randomisation part J
  Interventions: Drug: Sotrovimab
- Molnupiravir (Active Comparator): First (main) randomisation part K
  [This arm is now closed to recruitment]
  Interventions: Drug: Molnupiravir
- Paxlovid (Active Comparator): First (main) randomisation part L
  [This arm is now closed to recruitment]
  Interventions: Drug: Paxlovid
- Baloxavir marboxil (Active Comparator): Randomisation part G (influenza)
  Interventions: Drug: Baloxavir Marboxil
- Oseltamivir (Active Comparator): Randomisation part H (influenza)
  Interventions: Drug: Oseltamivir
- Low-dose corticosteroids: Dexamethasone (influenza arm) (Active Comparator): Randomisation part I (influenza)
  Interventions: Drug: Low-dose corticosteroids: Dexamethasone
- Low-dose corticosteroids: Dexamethasone (pneumonia arm) (Active Comparator): Randomisation part M (community-acquired pneumonia)
  Interventions: Drug: Low-dose corticosteroids: Dexamethasone

INTERVENTIONS:
Drug: Lopinavir-Ritonavir — Lopinavir 400mg-Ritonavir 100mg by mouth (or nasogastric tube) every 12 hours for 10 days.
  Arms: Lopinavir-Ritonavir
Drug: Corticosteroid — Corticosteroid in the form of dexamethasone administered as an oral (liquid or tablets) or intravenous preparation 6 mg once daily for 10 days. In pregnancy or breastfeeding women, prednisolone 40 mg administered by mouth (or intravenous hydrocortisone 80 mg twice daily) should be used instead of dexamethasone. Corticosteroid (in children ≤44 weeks gestational age, or >44 weeks gestational age with PIMS-TS only) in the form of Hydrocortisone or Methylprednisolone sodium succinate (see Protocol for timing and dosage)
  Arms: Low dose corticosteroids
Drug: Hydroxychloroquine — Hydroxychloroquine by mouth for a total of 10 days (see Protocol for timing and dosage).
  Arms: Hydroxychloroquine
Drug: Azithromycin — Azithromycin 500mg by mouth (or nasogastric tube) or intravenously once daily for 10 days.
  Arms: Azithromycin
Biological: Convalescent plasma — Single unit of ABO compatible convalescent plasma (275mls +/- 75 mls) intravenous per day on study days 1 (as soon as possible after randomisation) and 2 (with a minimum of 12 hour interval between 1st and 2nd units).
  Arms: Convalescent plasma
Drug: Tocilizumab — Tocilizumab by intravenous infusion with the dose determined by body weight (see Protocol for dosage)
  Arms: Tocilizumab
Biological: Immunoglobulin — Intravenous immunoglobulin (IVIg) for children >44 weeks gestational age and <18 years with PIMS-TS only (see Protocol for dosage)
  Arms: Intravenous Immunoglobulin
Drug: Synthetic neutralising antibodies — Patients ≥12 years only with COVID-19 pneumonia: A single dose of REGN10933 + REGN10987 8 g (4 g of each monoclonal antibody) in 250ml 0.9% saline infused intravenously over 60 minutes +/- 15 minutes as soon as possible after randomisation
  Other Names: REGEN-COV; casirivimab and imdevimab
  Arms: Synthetic neutralising antibodies
Drug: Aspirin — 150 mg by mouth (or nasogastric tube) or per rectum once daily until discharge, for adults ≥18 years old.
  Arms: Aspirin
Drug: Colchicine — 1 mg after randomisation followed by 500mcg 12 hours later and then 500 mcg twice daily by mouth or nasogastric tube for 10 days in total, for men ≥18 years old and women ≥55 years old only
  Arms: Colchicine
Drug: Baricitinib — UK [age ≥2 years with COVID pneumonia] and India [age ≥18 years with COVID-19 pneumonia]: 4 mg once daily by mouth or nasogastric tube for 10 days in total.
  Arms: Baricitinib
Drug: Anakinra — For children ≥1 <18 years old only: subcutaneously or intravenously once daily for 7 days or discharge (if sooner). NB Anakinra will be excluded from the randomisation of children <10 kg in weight.
  Arms: Anakinra
Drug: Dimethyl fumarate — Early phase assessment. UK adults ≥18 years old only (excluding those on ECMO). 120 mg every 12 hours for 4 doses followed by 240 mg every 12 hours by mouth for 8 days (10 days in total).
  Arms: Dimethyl fumarate
Drug: High Dose Corticosteroid — Adults ≥18 years old with hypoxia only. Dexamethasone 20 mg (base) once daily by mouth, nasogastric tube or intravenous infusion for 5 days follow by dexamethasone 10 mg (base) once daily by mouth, nasogastric tube or intravenous infusion for 5 days.
  Arms: High Dose Corticosteroids
Drug: Empagliflozin — Adults ≥18 years old only. 10 mg once daily by mouth for 28 days (or until discharge, if earlier).
  Arms: Empagliflozin
Drug: Sotrovimab — UK patients ≥12 years old. 1000 mg in 100 mL 0.9% sodium chloride or 5% dextrose by intravenous infusion over 1 hour as soon as possible after randomisation.
  Arms: Sotrovimab
Drug: Molnupiravir — Patients ≥18 years old. 800 mg twice daily for 5 days by mouth.
  Arms: Molnupiravir
Drug: Paxlovid — UK patients ≥18 years old. 300/100 mg twice daily for 5 days by mouth.
  Other Names: nirmatrelvir/ritonavir
  Arms: Paxlovid
Drug: Baloxavir Marboxil — Patients ≥12 years old in the UK (or ≥18 years old in other countries), with or without SARS-CoV-2 co-infection.
  40mg (or 80mg if weight ≥80kg) once daily by mouth or nasogastic tube to be given on day 1 and day 4.
  Other Names: Xofluza
  Arms: Baloxavir marboxil
Drug: Oseltamivir — Any age in the UK (or ≥18 years old in other countries), with or without SARS-CoV-2 co-infection.
  75mg twice daily by mouth or nasogastric tube for five days. (See Protocol for detailed dosage information)
  Other Names: Tamiflu
  Arms: Oseltamivir
Drug: Low-dose corticosteroids: Dexamethasone — Any age in the UK (or ≥18 years old in other countries), without suspected or confirmed SARS-CoV-2 infection, and with clinical evidence of hypoxia (i.e. receiving oxygen or with oxygen saturations <92% on room air) 6mg once daily given orally or intravenously for ten days or until discharge (whichever happens earliest)
  Arms: Low-dose corticosteroids: Dexamethasone (influenza arm)
Drug: Low-dose corticosteroids: Dexamethasone — ≥18 years old) with a diagnosis of community-acquired pneumonia (with planned antibiotic use and without suspected or confirmed SARS-CoV-2, influenza, active pulmonary tuberculosis, or Pneumocystis jirovecii infection) 6mg once daily given orally or intravenously for ten days or until discharge (whichever happens earliest)
  Arms: Low-dose corticosteroids: Dexamethasone (pneumonia arm)

SUMMARY:
RECOVERY is a randomised trial of treatments to prevent death in patients hospitalised with pneumonia.

The treatments being investigated are:

COVID-19: Lopinavir-Ritonavir, Hydroxychloroquine, Corticosteroids, Azithromycin, Colchicine, IV Immunoglobulin (children only), Convalescent plasma, Casirivimab+Imdevimab, Tocilizumab, Aspirin, Baricitinib, Empagliflozin, Sotrovimab, Molnupiravir, Paxlovid or Anakinra (children only)

Influenza: Baloxavir marboxil, Oseltamivir, Low-dose corticosteroids - Dexamethasone

Community-acquired pneumonia: Low-dose corticosteroids - Dexamethasone

DETAILED DESCRIPTION:
The RECOVERY trial has already shown that:

* Dexamethasone (a type of steroid) reduces the risk of dying for patients hospitalised with COVID-19 receiving oxygen,
* Regeneron's monoclonal antibody combination reduces deaths for hospitalised COVID-19 patients who have not mounted their own immune response,
* Tocilizumab reduces the risk of death when given to hospitalised patients with severe COVID-19. It also shortens the time until patients are successfully discharged from hospital and reduces the need for a mechanical ventilator.
* Baricitinib reduces the risk of death when given to hospitalised patients with severe COVID-19.
* In patients hospitalised for COVID-19 with clinical hypoxia but requiring either no oxygen or simple oxygen only, higher dose corticosteroids significantly increased the risk of death compared to usual care, which included low dose corticosteroids.

The trial also concluded that there is no beneficial effect of hydroxychloroquine, lopinavir-ritonavir, azithromycin, convalescent plasma, colchicine, aspirin, dimethyl fumarate or empagliflozin in patients hospitalised with COVID-19, and these arms have been closed to recruitment.

BACKGROUND: In early 2020, as this protocol was being developed, there were no approved treatments for COVID-19, a disease induced by the novel coronavirus SARSCoV-2 that emerged in China in late 2019. The UK New and Emerging Respiratory Virus Threats Advisory Group (NERVTAG) advised that several possible treatments should be evaluated, including Lopinavir-Ritonavir, low-dose corticosteroids, and Hydroxychloroquine (which has now been done). A World Health Organization (WHO) expert group issued broadly similar advice. These groups also advised that other treatments will soon emerge that require evaluation.

Since then, progress in COVID-19 treatment has highlighted the need for better evidence for the treatment of pneumonia caused by other pathogens, such as influenza and bacteria, for which therapies are widely used without good evidence of benefit or safety.

ELIGIBILITY AND RANDOMISATION: This protocol (v27.0 as of Dec 2023) describes a randomised trial among patients hospitalised with pneumonia caused by COVID-19, influennza or other organisms. All eligible patients are randomly allocated between several treatment arms, each to be given in addition to the usual standard of care in the participating hospital. The study is subdivided into several parts, according to whether participants are children or adults, and by geographic area. The study is dynamic, and treatments are added and removed as results and suitable treatments become available. The parts in the current version of the protocol are as follows:

Part A (COVID-19): discontinued in Protocol v19.0, (children's recruitment to Part A discontinued in Protocol v17.1)

Part B (COVID-19): discontinued in Protocol v16.0.

Part C (COVID-19): discontinued in Protocol v15.0.

Part D (COVID-19): discontinued in Protocol v20.0

Part E (COVID-19): Adults ≥18 years old with hypoxia only, randomised to high-dose corticosteroids vs no additional treatment.

Part F (COVID-19): discontinued in Protocol v26.0

Part G (Influenza): UK patients ≥12 years old (≥18 years old in other countries), with or without SARS-CoV-2 co-infection, randomised to baloxavir marboxil vrs no additional treatment

Part H (Influenza): UK patients ≥12 years old (≥18 years old in other countries), with or without SARS-CoV-2 co-infection, randomised to oseltamivir vrs no additional treatment

Part I (Influenza): UK patients any age (≥18 years old in other countries), without suspected or confirmed SARS-CoV-2 infection, and with clinical evidence of hypoxia (i.e. receiving oxygen or with oxygen saturations <92% on room air), randomised to Low-dose corticosteroids: Dexamethasone vrs no additional treatment.

Part J (COVID-19): UK patients ≥12 years old, randomised to sotrovimab vs no additional treatment.

Park K (COVID-19): discontinued in Protocol v26.0

Park L (COVID-19): discontinued in Protocol v26.0

Part M (Community-acquired pneumonia with planned antibiotic treatment and without suspected or confirmed SARS-CoV-2, influenza, active pulmonary tuberculosis, or Pneumocystis pneumonia): Patients ≥18 years old randomised to Low-dose corticosteroids: Dexamethasone vs no additional treatment.

Children with PIMS-TS: Tocilizumab vs anakinra vs no additional treatment (UK only) (discontinued in Protocol v23.1).

For patients for whom not all the trial arms are appropriate or at locations where not all are available, randomisation will be between fewer arms.

ADAPTIVE DESIGN: The interim trial results will be monitored by an independent Data Monitoring Committee (DMC). The most important task for the DMC will be to assess whether the randomised comparisons in the study have provided evidence on mortality that is strong enough (with a range of uncertainty around the results that is narrow enough) to affect national and global treatment strategies. In such a circumstance, the DMC will inform the Trial Steering Committee who will make the results available to the public and amend the trial arms accordingly. New trial arms can be added as evidence emerges that other candidate therapeutics should be evaluated.

OUTCOMES: The main outcomes will be death, discharge, need for ventilation and need for renal replacement therapy. For the main analyses, follow-up will be censored at 28 days after randomisation. Additional information on longer term outcomes may be collected through review of medical records or linkage to medical databases where available (such as those managed by NHS Digital and equivalent organisations in the devolved nations).

SIMPLICITY OF PROCEDURES: To facilitate collaboration, even in hospitals that suddenly become overloaded, patient enrolment (via the internet) and all other trial procedures are greatly streamlined. Informed consent is simple and data entry is minimal. Randomisation via the internet is simple and quick, at the end of which the allocated treatment is displayed on the screen and can be printed or downloaded. Key follow-up information is recorded at a single timepoint and may be ascertained by contacting participants in person, by phone or electronically, or by review of medical records and databases.

DATA TO BE RECORDED: At randomisation, information will be collected on the identity of the randomising clinician and of the patient, age, sex, major co-morbidity, pregnancy, COVID-19 onset date and severity, and any contraindications to the study treatments. The main outcomes will be death (with date and probable cause), discharge (with date), need for ventilation (with number of days recorded) and need for renal replacement therapy. Reminders will be sent if outcome data have not been recorded by 28 days after randomisation. Suspected Unexpected Serious Adverse Reactions (SUSARs) to one of the study medication (eg, Stevens-Johnson syndrome, anaphylaxis, aplastic anaemia) will be collected and reported in an expedited fashion. Other adverse events will not be recorded but may be available through linkage to medical databases.

NUMBERS TO BE RANDOMISED: The larger the number randomised the more accurate the results will be, but the numbers that can be randomised will depend critically on how large the epidemic becomes. If substantial numbers are hospitalised in the participating centres then it may be possible to randomise several thousand with mild disease and a few thousand with severe disease, but realistic, appropriate sample sizes could not be estimated at the start of the trial.

HETEROGENEITY BETWEEN POPULATIONS: If sufficient numbers are studied, it may be possible to generate reliable evidence in certain patient groups (e.g. those with major comorbidity or who are older). To this end, data from this study may be combined with data from other trials of treatments for COVID-19, such as those being planned by the WHO.

ADD-ON STUDIES: Particular countries or groups of hospitals, may well want to collaborate in adding further measurements or observations, such as serial virology, serial blood gases or chemistry, serial lung imaging, or serial documentation of other aspects of disease status. While well-organised additional research studies of the natural history of the disease or of the effects of the trial treatments could well be valuable (although the lack of placebo control may bias the assessment of subjective side-effects, such as gastrointestinal problems), they are not core requirements.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for the study if all of the following are true:

(i) Hospitalised

(ii) Pneumonia syndrome

In general, pneumonia should be suspected when a patient presents with:

1. typical symptoms of a new respiratory tract infection (e.g. influenza-like illness with fever and muscle pain, or respiratory illness with cough and shortness of breath); and
2. objective evidence of acute lung disease (e.g. consolidation or ground-glass shadowing on X-ray or CT, hypoxia, or compatible clinical examination); and
3. alternative causes have been considered unlikely or excluded (e.g. heart failure).

However, the diagnosis remains a clinical one based on the opinion of the managing doctor (the above criteria are just a guide).

(iii) One of the following diagnoses:

1. Confirmed SARS-CoV-2 infection (including patients with influenza co-infection)
2. Confirmed influenza A or B infection (including patients with SARS-CoV-2 co-infection)
3. Community-acquired pneumonia with planned antibiotic treatment (excluding patients with suspected or confirmed SARS-CoV-2, influenza, active pulmonary tuberculosis or Pneumocystis jirovecii pneumonia)

Exclusion criteria:

(iv) No medical history that might, in the opinion of the attending clinician, put the patient at significant risk if he/she were to participate in the trial

Participants will be excluded if the attending clinician believes that there is a specific contra-indication to one of the active drug treatment arms (see Protocol Appendix 2; section 8.2, and Appendix 3; section 8.3 for children, and Appendix 4 for pregnant and breastfeeding women), or that the patient should definitely be receiving one of the active drug treatment arms then that arm will not be available for randomisation for that patient. For patients who lack capacity, an advanced directive or behaviour that clearly indicates that they would not wish to participate in the trial would be considered sufficient reason to exclude them from the trial.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70000 (Estimated)
Dates: Start 2020-03-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2036-06-30 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | Within 28 days after randomisation
  For each pairwise comparison with the 'no additional treatment' arm, the primary objective is to provide reliable estimates of the effect of study treatments on all-cause mortality.
Influenza co-primary outcome: All-cause mortality (with subsidiary analysis of cause of death and death at various timepoints following discharge) | Within 28 days after randomisation
Influenza co-primary outcome: Time to discharge alive from hospital | Within the first 28-days

SECONDARY OUTCOMES:
COVID-19 & community-acquired pneumonia: Duration of hospital stay | Within 28 days and up to 6 months after the main randomisation
  To assess the effects of study treatment on number of days stay in hospital
COVID-19 & community-acquired pneumonia: Composite endpoint of death or need for mechanical ventilation or ECMO | Within 28 days and up to 6 months after the main randomisation
  Among patients not on invasive mechanical ventilation at baseline, the number of patients with a composite endpoint of death or need for invasive mechanical ventilation or ECMO.
Influenza: Composite endpoint of death or need for mechanical ventilation or ECMO | Within 28 days and up to 6 months after the main randomisation
  Among patients not on invasive mechanical ventilation at baseline, the number of patients with a composite endpoint of death or need for invasive mechanical ventilation or ECMO.

OTHER OUTCOMES:
Need for (and duration of) ventilation | Within 28 days and up to 6 months after the main randomisation
  To assess the effects of study treatment on number of patients who needed any ventilation and (for invasive mechanical ventilation) the number of days it was required
Need for renal replacement | Within 28 days and up to 6 months after the main randomisation
  To assess the effects of study treatment on number of patients who needed renal replacement therapy
Number of patients who had thrombotic events | Within 28 days and up to 6 months after the main randomisation
  To assess the effects of study treatment on number of patients who had thrombotic events, defined as either (i) acute pulmonary embolism; (ii) deep vein thrombosis; (iii) ischaemic stroke; (iv) myocardial infarction; or (v) systemic arterial embolism.

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Horby, Principal Investigator — University of Oxford
Locations (7):
- Kumasi Center for Collaborative Research in Tropical Medicine KNUST, Kumasi, Ghana
- Indian Council of Medical Research, Division of Epidemiology and Communicable Diseases, New Delhi, India
- Eijkman Oxford Clinical Research Unit (EOCRU), Eijkman Institute for Molecular Biology, Jakarta, Indonesia
- Clinical Trial Unit, Oxford University Clinical Research Unit-Nepal, Patan Academy of Health Sciences, Kathmandu, Nepal
- Wits Health Consortium, Johannesburg, South Africa
- Nuffield Department of Population Health, University of Oxford, Oxford, United Kingdom
- Oxford University Clinical Research Unit, Centre for Tropical Medicine, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
RECOVERY data will be made available via the Infectious Diseases Data Observatory (IDDO). Researchers will be able to apply via the IDDO Data Access process - https://www.iddo.org/covid19/data-sharing/accessing-data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: It is anticipated that some datasets will be available by Q1/2024.
Access Criteria: RECOVERY data will be made available via the Infectious Diseases Data Observatory (IDDO). Researchers will be able to apply via the IDDO Data Access process.
URL: https://www.iddo.org/covid19/data-sharing/accessing-data

REFERENCES:
- [Result] RECOVERY Collaborative Group; Horby P, Lim WS, Emberson JR, Mafham M, Bell JL, Linsell L, Staplin N, Brightling C, Ustianowski A, Elmahi E, Prudon B, Green C, Felton T, Chadwick D, Rege K, Fegan C, Chappell LC, Faust SN, Jaki T, Jeffery K, Montgomery A, Rowan K, Juszczak E, Baillie JK, Haynes R, Landray MJ. Dexamethasone in Hospitalized Patients with Covid-19. N Engl J Med. 2021 Feb 25;384(8):693-704. doi: 10.1056/NEJMoa2021436. Epub 2020 Jul 17. PMID 32678530
- [Result] RECOVERY Collaborative Group. Lopinavir-ritonavir in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet. 2020 Oct 24;396(10259):1345-1352. doi: 10.1016/S0140-6736(20)32013-4. Epub 2020 Oct 5. PMID 33031764
- [Result] RECOVERY Collaborative Group; Horby P, Mafham M, Linsell L, Bell JL, Staplin N, Emberson JR, Wiselka M, Ustianowski A, Elmahi E, Prudon B, Whitehouse T, Felton T, Williams J, Faccenda J, Underwood J, Baillie JK, Chappell LC, Faust SN, Jaki T, Jeffery K, Lim WS, Montgomery A, Rowan K, Tarning J, Watson JA, White NJ, Juszczak E, Haynes R, Landray MJ. Effect of Hydroxychloroquine in Hospitalized Patients with Covid-19. N Engl J Med. 2020 Nov 19;383(21):2030-2040. doi: 10.1056/NEJMoa2022926. Epub 2020 Oct 8. PMID 33031652
- [Result] RECOVERY Collaborative Group. Azithromycin in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet. 2021 Feb 13;397(10274):605-612. doi: 10.1016/S0140-6736(21)00149-5. Epub 2021 Feb 2. PMID 33545096
- [Result] RECOVERY Collaborative Group. Tocilizumab in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet. 2021 May 1;397(10285):1637-1645. doi: 10.1016/S0140-6736(21)00676-0. PMID 33933206
- [Result] RECOVERY Collaborative Group. Convalescent plasma in patients admitted to hospital with COVID-19 (RECOVERY): a randomised controlled, open-label, platform trial. Lancet. 2021 May 29;397(10289):2049-2059. doi: 10.1016/S0140-6736(21)00897-7. Epub 2021 May 14. PMID 34000257
- [Result] RECOVERY Collaborative Group. Colchicine in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet Respir Med. 2021 Dec;9(12):1419-1426. doi: 10.1016/S2213-2600(21)00435-5. Epub 2021 Oct 18. PMID 34672950
- [Result] RECOVERY Collaborative Group. Aspirin in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet. 2022 Jan 8;399(10320):143-151. doi: 10.1016/S0140-6736(21)01825-0. Epub 2021 Nov 17. PMID 34800427
- [Result] RECOVERY Collaborative Group. Casirivimab and imdevimab in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet. 2022 Feb 12;399(10325):665-676. doi: 10.1016/S0140-6736(22)00163-5. PMID 35151397
- [Result] RECOVERY Collaborative Group. Baricitinib in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial and updated meta-analysis. Lancet. 2022 Jul 30;400(10349):359-368. doi: 10.1016/S0140-6736(22)01109-6. PMID 35908569
- [Result] RECOVERY Collaborative Group. Dimethyl fumarate in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. medRxiv. 25 September 2022. doi.org/10.1101/2022.09.23.22280285
- [Result] RECOVERY Collaborative Group. Electronic address: recoverytrial@ndph.ox.ac.uk; RECOVERY Collaborative Group. Higher dose corticosteroids in patients admitted to hospital with COVID-19 who are hypoxic but not requiring ventilatory support (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet. 2023 May 6;401(10387):1499-1507. doi: 10.1016/S0140-6736(23)00510-X. Epub 2023 Apr 13. PMID 37060915
- [Result] RECOVERY Collaborative Group. Empagliflozin in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet Diabetes Endocrinol. 2023 Dec;11(12):905-914. doi: 10.1016/S2213-8587(23)00253-X. Epub 2023 Oct 18. PMID 37865101
- [Derived] RECOVERY Collaborative Group. Sotrovimab versus usual care in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet Infect Dis. 2026 Jan;26(1):34-45. doi: 10.1016/S1473-3099(25)00361-5. Epub 2025 Aug 28. PMID 40886716
- [Derived] RECOVERY Collaborative Group. Molnupiravir or nirmatrelvir-ritonavir plus usual care versus usual care alone in patients admitted to hospital with COVID-19 (RECOVERY): a randomised, controlled, open-label, platform trial. Lancet Infect Dis. 2025 Sep;25(9):1000-1010. doi: 10.1016/S1473-3099(25)00093-3. Epub 2025 May 15. PMID 40383127
- [Derived] RECOVERY Collaborative Group. Higher dose corticosteroids in hospitalised COVID-19 patients requiring ventilatory support (RECOVERY): a randomised, controlled, open-label, platform trial. EClinicalMedicine. 2025 Feb 12;81:103080. doi: 10.1016/j.eclinm.2025.103080. eCollection 2025 Mar. PMID 40036152
- [Derived] Pessoa-Amorim G, Goldacre R, Crichton C, Stevens W, Nunn M, King A, Murray D, Welsh R, Pinches H, Rees A, Morris EJA, Landray MJ, Haynes R, Horby P, Wallendszus K, Peto L, Campbell M, Harper C, Mafham M. Clinical trial results in context: comparison of baseline characteristics and outcomes of 38,510 RECOVERY trial participants versus a reference population of 346,271 people hospitalised with COVID-19 in England. Trials. 2024 Jun 29;25(1):429. doi: 10.1186/s13063-024-08273-9. PMID 38951929
- [Derived] RECOVERY Collaborative Group. Immunomodulatory therapy in children with paediatric inflammatory multisystem syndrome temporally associated with SARS-CoV-2 (PIMS-TS, MIS-C; RECOVERY): a randomised, controlled, open-label, platform trial. Lancet Child Adolesc Health. 2024 Mar;8(3):190-200. doi: 10.1016/S2352-4642(23)00316-4. Epub 2024 Jan 22. PMID 38272046
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Chevret S, Timsit JF, Biard L. Challenges of using external data in clinical trials- an illustration in patients with COVID-19. BMC Med Res Methodol. 2022 Dec 15;22(1):321. doi: 10.1186/s12874-022-01769-5. PMID 36522698
- [Derived] Hirsch C, Park YS, Piechotta V, Chai KL, Estcourt LJ, Monsef I, Salomon S, Wood EM, So-Osman C, McQuilten Z, Spinner CD, Malin JJ, Stegemann M, Skoetz N, Kreuzberger N. SARS-CoV-2-neutralising monoclonal antibodies to prevent COVID-19. Cochrane Database Syst Rev. 2022 Jun 17;6(6):CD014945. doi: 10.1002/14651858.CD014945.pub2. PMID 35713300
- [Derived] Kramer A, Prinz C, Fichtner F, Fischer AL, Thieme V, Grundeis F, Spagl M, Seeber C, Piechotta V, Metzendorf MI, Golinski M, Moerer O, Stephani C, Mikolajewska A, Kluge S, Stegemann M, Laudi S, Skoetz N. Janus kinase inhibitors for the treatment of COVID-19. Cochrane Database Syst Rev. 2022 Jun 13;6(6):CD015209. doi: 10.1002/14651858.CD015209. PMID 35695334
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Tume LN, Menzies JC, Ray S, Scholefield BR; UK Paediatric Intensive Care Society Study Group. Research Priorities for U.K. Pediatric Critical Care in 2019: Healthcare Professionals' and Parents' Perspectives. Pediatr Crit Care Med. 2021 May 1;22(5):e294-e301. doi: 10.1097/PCC.0000000000002647. PMID 33394942
- See also: RECOVERY Trial website (preliminary results, the Protocol, the Statistical Analysis Plan, and other trial documents can be downloaded from this website) — https://www.recoverytrial.net/